CLINICAL TRIAL: NCT05100355
Title: Management of the Lack of Blood Return on a Central Venous Catheter (CVC) Before Chemotherapy in a Day Unit: Phase III Randomised Multicentre Study
Brief Title: Management of the Lack of Blood Return on a Central Venous Catheter (CVC) Before Chemotherapy
Acronym: CATAREV-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: PHRC-I (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2021-07
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Catheter Dysfunction
Keywords: lack of CVC blood return; Central Venous Catheter (CVC); Day unit; Opacification; Contrast media; Medico-economic evaluation; Physiological serum; Chest X-ray
MeSH Terms: interventions — Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opacification (Active Comparator): Contrast agent injection
  Interventions: Procedure: Contrast agent injection
- Physiological serum injection (Experimental): Physiological serum injection
  Interventions: Procedure: Physiological serum injection

INTERVENTIONS:
Procedure: Physiological serum injection — In case of lack of CVC blood return, Physiological serum is injected in the CVC after Chest X-Ray
  Arms: Physiological serum injection
Procedure: Contrast agent injection — In case of lack of CVC blood return, Contrast agent is injected in the CVC after Chest X-Ray
  Arms: Opacification

SUMMARY:
Compare two methods of managing the lack of CVC blood return : opacification using contrast media injection or radio-clinical method with a simple chest X-ray followed by a rapid infusion of physiological serum

DETAILED DESCRIPTION:
The use of CVC is part of daily life in onco-hematology, particularly for chemotherapy treatments in the Day Unit (DU). Among the possible complications and dysfunctions, the most frequent is the lack of CVC blood return, which can be responsible for a disorganization of the patient's management in the Day Unit (delay in patient management).

In this study, the 2 most commonly used schemes are compared in a randomised multicentre study.

The first scheme is a radiological circuit with opacification using contrast media injection.

The second scheme is radio-clinical with a chest X-ray to check the correct functioning of the CVC followed by a rapid infusion of physiological serum.

The patient management is compared for the two schemes in term of delay (delay from start to end time of patient management). The safety and the cost of both schemes is compared.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, Age ≥ 18 years at time of study entry.
* Undergoing systemic chemotherapy on a CVC. Immunotherapy and targeted therapies are among the systemic therapies that are authorised
* Having already received at least one administration of treatment without difficulty.
* Coming for a new administration of treatment authorised by the usual biological assessment.
* First episode of lack of CVC blood return despite the usual positioning and injection- aspiration manoeuvres
* No abnormality on inspection or palpation (turning) of the CVC.
* Patient has valid health insurance.
* Patient information and signature of informed consent.

Exclusion Criteria:

* Previous episode of lack of CVC blood return whether explored or not.
* Patient currently treated in an interventional therapeutic trial.
* Patient with a Picc-line implantable device.
* Suspected CVC infection or thrombosis.
* Planned chemotherapy with vesicant agent (anthracyclines).
* Possible CVC disjunction.
* Allergy to X-ray contrast agent or creatinine clearance below 30ml/min prohibiting an iodine injection.
* Pregnant, likely to be pregnant or breastfeeding woman.
* Persons deprived of their liberty, under a measure of safeguard of justice, under guardianship or placed under the authority of a guardian.
* Impossibility of undergoing medical monitoring of the trial for geographical, social or psychological reasons, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Compare the delay between randomisation (determination of the lack of blood return) and the decision to initiate or not the chemotherapy protocol on the same day, for both procedures | 1 day
  Time between randomisation and the decision to initiate or not the chemotherapy

SECONDARY OUTCOMES:
Medico-economic evaluation of both procedures | 3 months
  Average cost of the patient management for each procedure
Medico-economic evaluation of both procedures | 3 months
  Number of new lack of catheter blood return events
Medico-economic evaluation of both procedures | 3 months
  Number of complications events
Evaluate the frequency of recurrence of lack of CVC blood return | 3 months
  Number of new events of lack of CVC blood return
Evaluate the frequency of recurrence of new re-opacification events | 3 months
  Number of new CVC re-opacification events
Evaluate the frequency of CVC replacement | 3 months
  Number of new catheter replacements
Quantify systemic CVC infectious complications | 14 days
  Number of Systemic CVC infectious complications
Assess allergic reactions | 24 hours
  Number of Allergic reactions requiring at least oral therapy
Assess renal impairment | 28 days
  Increase in creatinine to > 1.5 times the most recent screening value
Assess the treatment delay due to CVC blood return | 1 day
  Number of CVC blood return that led to delay the treatment to the day after

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut du Cancer Sainte Catherine Avignon Provence, Avignon
  - Ch Cholet, Cholet
  - CHD La Roche Sur yon, La Roche-sur-Yon
  - Centre Eugène Marquis, Rennes
  - CH Yves Le Foll, Saint-Brieuc
  - Audrey ROLLOT, Saint-Herblain
  - Centre Hospitalier de St Malo, St-Malo
  - CHBA Vannes, Vannes